CLINICAL TRIAL: NCT05752981
Title: Full-head Coverage Multi-channel Time-resolved Functional Near Infrared Spectroscopy for Early Detection and Prevention of Perioperative Brain Injury
Brief Title: Multi-channel Time-resolved Functional Near Infrared Spectroscopy for Prevention of Perioperative Brain Injury
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Jason Chui, Anesthesiologist, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: tr-fNIRS
Record Dates: First submitted 2023-02-02; First posted 2023-03-03 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Cerebral Oxygenation
Keywords: neuromonitoring; cerebral oxygenation; stroke; anesthesia
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- tr-FNIRS neuromonitor: During shoulder surgery, the tr-fNIRS (time-resolved (tr) functional near infrared spectroscopy (fNIRS) (tr-fNIRS)) neuromonitor will be used to gather data on cerebral oxygenation of multiple brain regions for these patients. No intervention will be administered based on the results of the tr-fNIRS.
  Interventions: Device: multichannel time-resolved (tr) functional near infrared spectroscopy (fNIRS) (tr-fNIRS)

INTERVENTIONS:
Device: multichannel time-resolved (tr) functional near infrared spectroscopy (fNIRS) (tr-fNIRS) — Participants will be monitored during surgery using the multichannel time-resolved (tr) functional near infrared spectroscopy (fNIRS) (tr-fNIRS). This study is observational in nature and no intervention will be applied based on the results of the tr-fNIRS device.

SUMMARY:
Covert stroke occurs in one out of fourteen patients during or shortly after surgery, and may result in long-term disability. Fortunately, stroke that occurs during non-cardiac surgery is most commonly caused by inadequate blood flow to the brain and is, therefore, preventable if it can be detected early. Current clinical tools used to monitor the brain during surgery do not have the accuracy nor the spatial coverage - they only monitor one small region of the brain. In this study, the investigators plan to apply a cutting-edge optical device, tr-fNIRS, to monitor the whole brain during shoulder surgery. The primary aim is to determine any regional differences in cerebral oxygenation (ScO2) and cerebral autoregulation (CA)between brain regions during surgery and especially during various physiological challenges, such as hypotension. The investigators hypothesize that certain brain regions are more likely to develop cerebral desaturation and impaired CA, and are more prone to brain injury than the frontal lobe region which is the traditional monitoring site. The investigators also hypothesize that cerebral desaturation (or hypoxic injury) events correlate with adverse postoperative neurological outcomes such as covert stroke, overt stroke and/or postoperative delirium.

DETAILED DESCRIPTION:
Perioperative stroke is a significant complication after surgery. Unfortunately, covert stroke occurs in one out of fourteen elderly patients after non-cardiac surgery and is associated with an increased risk of long-term cognitive decline. Further, perioperative overt stroke is associated with an 8-fold increase in perioperative mortality, prolonged length of hospital stay, and decreased quality of life. For shoulder surgery performed in the beach chair position, due to systemic hypotension and reduction in cerebral perfusion pressure, cerebral desaturation events and impaired cerebral autoregulation can occur in up to 80% of patients. Most perioperative stroke in non-cardiac surgery is ischemic and is related to brain hypoperfusion. Importantly, brain hypoperfusion is potentially modifiable with simple measures such as increasing systemic blood pressure (BP) if brain ischemia is identified early enough. However, deliberate hypertension is not devoid of risk and there is currently no effective monitor that can detect brain hypoperfusion during surgery.

Cerebral oxygenation has been used clinically as a measure of adequate brain perfusion during surgery. An early clinical trial at Western found that monitoring cerebral oxygenation was associated with fewer cases of major organ dysfunction in cardiac surgery patients. Despite this promising initial finding, current commercial cerebral oximeters have a number of limitations that prevent reliable perioperative neuromonitoring, including non-specificity due to signal contamination from extracerebral tissue, especially during administration of vasoconstrictors or hypothermia. In addition, current commercial cerebral oximeters only have two channels to monitor the frontal lobe regions (i.e., anterior cerebral artery territory). This monitoring strategy assumes that cerebral oxygenation is homogenous across different brain regions so that measurements from the frontal lobe regions can be used clinically to represent the adequacy of global brain oxygenation. Such a limited spatial coverage may result in undetected stroke, despite the patients having apparently normal cerebral oxygenation in the frontal regions throughout surgery. The current research project employs multi-channel tr-fNIRS to address these limitations, with the goal of timely detection and prevention of ischemic brain injury.

Multi-channel tr-fNIRS (time-resolved (tr) functional near infrared spectroscopy (fNIRS) (tr-fNIRS)) is an emerging brain-imaging technology that was originally developed to explore changes in cerebral oxygenation generated by cortical neuronal activity during various cognitive tasks such as speech, sensory and motor functions, and emotion. This is because tr-fNIRS can measure such subtle cerebral oxygenation changes in milliseconds (up to 100 ms) that accompany neuro-activation such as finger-tapping. The investigators has built several tr-fNIRS devices and have the expertise of adapting the full head coverage tr-fNIRS device to perioperative neuromonitoring. Furthermore, tr-fNIRS operate by sending short (picosecond) pulses of light into the head and precisely measures the time of travel of each photon in the tissue. Since there is an equivalence between time and distance, photons that are detected right after the pulse have only probed the extracerebral layers (scalp and skull) while photons that are detected long after (1-2 ms) the pulse have travelled deep into the brain tissues. The investigators have recently shown that this approach reduces the signal contaminations of the extracerebral layers from 80% with current commercial NIRS devices to less than 8% with tr-fNIRS. In this study, the investigators will employ a state-of-the-art full head coverage tr-fNIRS device to monitor the entire brain, as opposed to only select regions (such as the limited capabilities of the current cerebral oximeters) in the perioperative setting. Together with in-house analysis algorithms, the full head coverage tr-fNIRS can detect specific brain regions at-risk of ischemic injury with a high degree of certainty because of greater spatial resolution (in cm) and less signal contamination from extracerebral tissue.

All study participants will be recruited and consented adhering to the local ethics guidelines. For all study participants, the surgical and anesthetic management of the patients will be conducted in a standard fashion and will not be altered in this study. The exception is that tr-fNIRS will be used to monitor regional brain oxygenation from anesthesia induction to completion of surgery. The surgeons, anesthesiologists, and nurses will be blinded to the monitor/measurements during the procedure. No intervention will be administered based on the results of the tr-fNIRS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years old)
* Scheduled to have elective shoulder surgery in the beach-chair position under general anesthesia
* Provide informed consent

Exclusion Criteria:

i) have skin/scalp lesions that preclude the application of fNIRS device to the head ii) lack of written consent iii) emergency surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Shoulder surgery patients were chosen as the study population because of the high frequency of intraoperative hypotensive and cerebral desaturation events that may occur during this procedure, and the unique physiological changes such as impaired cerebral autoregulation that accompany the beach chair surgical positioning. This unique but commonly encountered operative condition create ischemic challenges and injury to the brain and provide opportunities to assess the spatial and temporal differences of cerebral desaturation patterns experienced during hypotensive and other physiological challenges, and to refine the tr-fNIRS device for perioperative applications.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of intraoperative hemodynamic parameter on regional differences in cerebral oxygenation (ScO2) between brain regions during surgery | Duration of surgical procedure
  cerebral oxygenation (ScO2) between brain regions will be done by assessing the data collected by the tr-fNIRS monitor during surgery.

SECONDARY OUTCOMES:
Regional differences in cerebral autoregulation in beach-chair position under general anesthesia as measured by the tr-fNIRS monitor (Hz) data outputs. | Duration of surgery
  Cerebral autoregulation index will be calculated based on the data collected by the tr-fNIRS monitor during surgery.
To assess the association between cerebral desaturation (or hypoxic injury) events in multiple brain regions to clinical outcomes such as stroke and delirium | Up to 72 hours following surgery or until discharge from hospital.
  Covert stroke will be assessed by performing a postoperative MRI. Neurological deficits will be assessed by physical examination and delirium will be assessed by 3D CAM administration).

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mrkobrada M, Hill MD, Chan MT, Sigamani A, Cowan D, Kurz A, Sessler DI, Jacka M, Graham M, Dasgupta M, Dunlop V, Emery DJ, Gulka I, Guyatt G, Heels-Ansdell D, Murkin J, Pettit S, Sahlas DJ, Sharma M, Sharma M, Srinathan S, St John P, Tsai S, Gelb AW, O'Donnell M, Siu D, Chiu PW, Sharath V, George A, Devereaux PJ. Covert stroke after non-cardiac surgery: a prospective cohort study. Br J Anaesth. 2016 Aug;117(2):191-7. doi: 10.1093/bja/aew179. PMID 27440630
- [Background] Mashour GA, Shanks AM, Kheterpal S. Perioperative stroke and associated mortality after noncardiac, nonneurologic surgery. Anesthesiology. 2011 Jun;114(6):1289-96. doi: 10.1097/ALN.0b013e318216e7f4. PMID 21478735
- [Background] NeuroVISION Investigators. Perioperative covert stroke in patients undergoing non-cardiac surgery (NeuroVISION): a prospective cohort study. Lancet. 2019 Sep 21;394(10203):1022-1029. doi: 10.1016/S0140-6736(19)31795-7. Epub 2019 Aug 15. PMID 31422895
- [Background] Salazar JD, Wityk RJ, Grega MA, Borowicz LM, Doty JR, Petrofski JA, Baumgartner WA. Stroke after cardiac surgery: short- and long-term outcomes. Ann Thorac Surg. 2001 Oct;72(4):1195-201; discussion 1201-2. doi: 10.1016/s0003-4975(01)02929-0. PMID 11603436
- [Background] McCulloch TJ, Liyanagama K, Petchell J. Relative hypotension in the beach-chair position: effects on middle cerebral artery blood velocity. Anaesth Intensive Care. 2010 May;38(3):486-91. doi: 10.1177/0310057X1003800312. PMID 20514957
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS, Vaughn J, Nisman M. Cerebral oxygen desaturation events assessed by near-infrared spectroscopy during shoulder arthroscopy in the beach chair and lateral decubitus positions. Anesth Analg. 2010 Aug;111(2):496-505. doi: 10.1213/ANE.0b013e3181e33bd9. Epub 2010 May 27. PMID 20508134
- [Background] Salazar D, Sears BW, Aghdasi B, Only A, Francois A, Tonino P, Marra G. Cerebral desaturation events during shoulder arthroscopy in the beach chair position: patient risk factors and neurocognitive effects. J Shoulder Elbow Surg. 2013 Sep;22(9):1228-35. doi: 10.1016/j.jse.2012.12.036. Epub 2013 Feb 15. PMID 23415820
- [Background] Lee JH, Min KT, Chun YM, Kim EJ, Choi SH. Effects of beach-chair position and induced hypotension on cerebral oxygen saturation in patients undergoing arthroscopic shoulder surgery. Arthroscopy. 2011 Jul;27(7):889-94. doi: 10.1016/j.arthro.2011.02.027. Epub 2011 May 28. PMID 21620637
- [Background] Sun LY, Chung AM, Farkouh ME, van Diepen S, Weinberger J, Bourke M, Ruel M. Defining an Intraoperative Hypotension Threshold in Association with Stroke in Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):440-447. doi: 10.1097/ALN.0000000000002298. PMID 29889106
- [Background] Joshi B, Ono M, Brown C, Brady K, Easley RB, Yenokyan G, Gottesman RF, Hogue CW. Predicting the limits of cerebral autoregulation during cardiopulmonary bypass. Anesth Analg. 2012 Mar;114(3):503-10. doi: 10.1213/ANE.0b013e31823d292a. Epub 2011 Nov 21. PMID 22104067
- [Background] Ono M, Joshi B, Brady K, Easley RB, Zheng Y, Brown C, Baumgartner W, Hogue CW. Risks for impaired cerebral autoregulation during cardiopulmonary bypass and postoperative stroke. Br J Anaesth. 2012 Sep;109(3):391-8. doi: 10.1093/bja/aes148. Epub 2012 Jun 1. PMID 22661748
- [Background] Brady KM, Hudson A, Hood R, DeCaria B, Lewis C, Hogue CW. Personalizing the Definition of Hypotension to Protect the Brain. Anesthesiology. 2020 Jan;132(1):170-179. doi: 10.1097/ALN.0000000000003005. No abstract available. PMID 31644437
- [Background] Lee JM, Grabb MC, Zipfel GJ, Choi DW. Brain tissue responses to ischemia. J Clin Invest. 2000 Sep;106(6):723-31. doi: 10.1172/JCI11003. No abstract available. PMID 10995780
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Grocott HP, Davie SN. Future uncertainties in the development of clinical cerebral oximetry. Front Physiol. 2013 Dec 18;4:360. doi: 10.3389/fphys.2013.00360. eCollection 2013. No abstract available. PMID 24385967
- [Background] Ogoh S, Sato K, Okazaki K, Miyamoto T, Secher F, Sorensen H, Rasmussen P, Secher NH. A decrease in spatially resolved near-infrared spectroscopy-determined frontal lobe tissue oxygenation by phenylephrine reflects reduced skin blood flow. Anesth Analg. 2014 Apr;118(4):823-9. doi: 10.1213/ANE.0000000000000145. PMID 24651237
- [Background] Erdoes G, Rummel C, Basciani RM, Verma R, Carrel T, Banz Y, Eberle B, Schroth G. Limitations of Current Near-Infrared Spectroscopy Configuration in Detecting Focal Cerebral Ischemia During Cardiac Surgery: An Observational Case-Series Study. Artif Organs. 2018 Oct;42(10):1001-1009. doi: 10.1111/aor.13150. Epub 2018 May 3. PMID 29726003
- [Background] Ban HY, Barrett GM, Borisevich A, Chaturvedi A, Dahle JL, Dehghani H, Dubois J, Field RM, Gopalakrishnan V, Gundran A, Henninger M, Ho WC, Hughes HD, Jin R, Kates-Harbeck J, Landy T, Leggiero M, Lerner G, Aghajan ZM, Moon M, Olvera I, Park S, Patel MJ, Perdue KL, Siepser B, Sorgenfrei S, Sun N, Szczepanski V, Zhang M, Zhu Z. Kernel Flow: a high channel count scalable time-domain functional near-infrared spectroscopy system. J Biomed Opt. 2022 Jan;27(7):074710. doi: 10.1117/1.JBO.27.7.074710. PMID 35043610
- [Background] Milej D, Shahid M, Abdalmalak A, Rajaram A, Diop M, St Lawrence K. Characterizing dynamic cerebral vascular reactivity using a hybrid system combining time-resolved near-infrared and diffuse correlation spectroscopy. Biomed Opt Express. 2020 Jul 23;11(8):4571-4585. doi: 10.1364/BOE.392113. eCollection 2020 Aug 1. PMID 32923065
- [Background] Milej D, Abdalmalak A, McLachlan P, Diop M, Liebert A, St Lawrence K. Subtraction-based approach for enhancing the depth sensitivity of time-resolved NIRS. Biomed Opt Express. 2016 Oct 7;7(11):4514-4526. doi: 10.1364/BOE.7.004514. eCollection 2016 Nov 1. PMID 27895992